CLINICAL TRIAL: NCT00698191
Title: Phase I/IIa: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells Transplantation For Refractory Systemic Lupus Erythematosus
Brief Title: Mesenchymal Stem Cells Transplantation for Refractory Systemic Lupus Erythematosus (SLE)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sun, Lingyun/ Prof., Nanjing University Medical College Affiliated Drum Tower Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSFC30772014
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Refractory Systemic Lupus Erythematosus
Keywords: Lupus Erythematosus,Systemic; Lupus Nephritis; Mesenchymal Stem Cells; Transplantation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Allogeneic MSC (AlloMSC)

INTERVENTIONS:
Biological: Allogeneic MSC (AlloMSC) — Intervention:
  Cyclophosphamide will be administered intravenously at at total dose of 0.8-1.8g 24 hours before transplantation.
  Allogeneic bone marrow derived mesenchymal stem cells (matched family donors)will be infused intravenously at 106 cells/kg body weight

SUMMARY:
This study will explore a new approach to treat patients with a medical condition known as systemic lupus erythematosus (SLE) who have been resistant to previous treatments using a new population of cells with capability to restore a normal immune system that will no longer attack the body.

The stated hypothesis is that the SLE condition is caused by an abnormal immune system that can be restored by replenishing the body with a new population of progenitor cells.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of allogeneic bone marrow derived mesenchymal stem cell (AlloMSC) transplantation in patients with refractory SLE. Patients with Lupus nephritis and refractory to corticosteroid or cyclophosphamide trials will be enrolled in this trial. The treatment intervention includes a 24 hour pretreatment with cyclophosphamide followed by AlloMSC transplantation. Patients will be admitted to the in-patient service for the 3-5 days for the transplant treatment and will be followed up in the outpatient clinic. All baseline lupus serology, renal function panels will be obtained at pre-treatment admission. Post-transplantation follow-up visits will be at monthly intervals for lupus serology and renal function tests, and every 3 months for analysis of T regulatory population. The transplanted patients will be evaluated by an integrated team of rheumatologists, hematologists and bone marrow transplant specialists every month for the entire duration of the trial (2 years) and every 6-12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the American College of Rheumatology (ACR) criteria of SLE, man or woman aged from 15 to 70 years old, SLEDAI≥8;
* Lupus nephritis with 24h urine protein≥1g;
* Refractory disease as determined by failure of the following regimens:

  * Trial of corticosteroids (oral prednisone more than 20 mg/day);
  * Trial of cyclophosphamide 0.4 ~ 0.6 / m2 every two weeks for six months, or other immunosuppressive drugs, such as MMF 2 g / day, for three months;
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital;
* Willing to use contraception throughout the study and for 12 mos following treatment.

Exclusion Criteria:

* Abnormal liver function (ALT higher than 3 times the normal value);
* End-stage renal failure;
* Severe heart and pulmonary failure, or other important organs damage;
* Undercontrolled infections
* Pregnant or breast feeding women, male or female who intended to recent pregnancy.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | Monthly
Lupus serology (ANA, dsDNA, C3, C4) | Monthly
Renal function (GFR, BUN, urinalysis) | Monthly

SECONDARY OUTCOMES:
Percentage of systemic T regulatory population | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Sun, M.D., Study Director — Nanjing University Medical College Affiliated Drum Tower Hospital
Locations (1):
- Department of Rheumatology and Immunology, Nanjing University Medical College Affiliated Drum Tower Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Jiang B, Sun L, Hao S, Li X, Xu Y, Hou Y. Estrogen modulates bone marrow-derived DCs in SLE murine model-(NZB x NZW) F1 female mice. Immunol Invest. 2008;37(3):227-43. doi: 10.1080/08820130801973328. PMID 18389442
- [Background] Jiang B, Sun L, Hao S, Li X, Hou Y. Estrogen distinctively modulates spleen DC from (NZB x NZW) F1 female mice in various disease development stages. Cell Immunol. 2007 Aug;248(2):95-102. doi: 10.1016/j.cellimm.2007.10.004. Epub 2007 Dec 3. PMID 18061155
- [Background] Sun LY, Zhang HY, Feng XB, Hou YY, Lu LW, Fan LM. Abnormality of bone marrow-derived mesenchymal stem cells in patients with systemic lupus erythematosus. Lupus. 2007;16(2):121-8. doi: 10.1177/0961203306075793. PMID 17402368
- [Derived] Liang J, Zhang H, Kong W, Deng W, Wang D, Feng X, Zhao C, Hua B, Wang H, Sun L. Safety analysis in patients with autoimmune disease receiving allogeneic mesenchymal stem cells infusion: a long-term retrospective study. Stem Cell Res Ther. 2018 Nov 14;9(1):312. doi: 10.1186/s13287-018-1053-4. PMID 30428931